CLINICAL TRIAL: NCT03380325
Title: The Effects of Iloprost Infusion on Capillary Recruitment and Whole-body Glucose Uptake in Type 2 Diabetic Patients - a Cross-over Trial.
Brief Title: The Effect of Iloprost on Capillary Recruitment and Insulin Sensitivity in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Erik Serne, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Bootcamp1
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Sensitivity/Resistance
Keywords: Capillary recruitment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

ARMS (2):
- Iloprost first (Experimental): Cross-over starts with iloprost intervention, then second clamp without iloprost.
  Interventions: Drug: Iloprost infusion
- Iloprost second (Experimental): Cross-over starts without iloprost intervention, then second clamp with iloprost.
  Interventions: Drug: Iloprost infusion

INTERVENTIONS:
Drug: Iloprost infusion — Iloprost is a stable prostacyclin analogue

SUMMARY:
This study examines the effects of iloprost - a stable prostacyclin analogue - on insulin-mediated muscle capillary recruitment and whole-body glucose uptake in a cross-over design.

DETAILED DESCRIPTION:
In type 2 diabetes impaired insulin-mediated muscle perfusion is thought to contribute to reduced whole-body glucose uptake. This study aims to identify iloprost - a stable prostacyclin analogue - as a possible therapeutic option to increase whole-body glucose uptake via enhancement of muscle perfusion.

All participants will be subjected to two hyperinsulinemic-euglycemic clamps; one with and one without simultaneous iloprost infusion in a randomized cross-over design. Microvascular blood volume will be measured by means of contrast-enhanced ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Male or female (post-menopausal)
* Age above 45 years and below 70 years
* BMI >30 kg/m2
* HbA1c < 80 mmol/mol or < 8,6% Subjects must use metformin
* Stable medication use
* Stable tension regulation (with or without medication)
* Subjects should be able to give informed consent

Exclusion Criteria:

* A history of cardiovascular event (Cerebrovascular event, myocardial infarction or pacemaker implantation)
* Severe-very severe lung emphysema (GOLD stage III-IV)
* Use of any antibiotics or proton pump inhibitor (PPI) in the past three months
* Use of any other antidiabetic medication besides metformin (e.g. SU-derivates, insulin)
* Use of a platelet inhibitor or cumarin derivate during
* Subjects participated in a lifestyle programme in the past 6 months (diet or exercise)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Rate of disappearance | During the clamp
  Glucose uptake in peripheral tissues during hyperinsulinemic euglycemic clamp
Capillary recruitment | Before and during the clamp
  Change in skeletal muscle en myocardial microvascular blood volume upon insulin infusion

SECONDARY OUTCOMES:
Continous cardiovascular monitoring | Before and during the clamp
  Diastolic blood pressure
Continous cardiovascular monitoring | Before and during the clamp
  Systolic blood pressure
Continous cardiovascular monitoring | Before and during the clamp
  Cardiac output
Continous cardiovascular monitoring | Before and during the clamp
  Heart rate
Continous cardiovascular monitoring | Before and during the clamp
  Stroke volume
Continous cardiovascular monitoring | Before and during the clamp
  Systemic vascular resistance

CONTACTS AND LOCATIONS:
Overall Officials: Erik Serné, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands